CLINICAL TRIAL: NCT02415309
Title: Premedication With Melatonin vs. Placebo in Patients Undergoing Interventional Pain Procedure
Brief Title: Premedication With Melatonin in Lumbar Medial Branch Block Procedure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Principal Investigator, Eugene Smith, LCDR, MD, United States Naval Medical Center, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NMCSD.2015.0048
Record Dates: First submitted 2015-04-06; First posted 2015-04-14 (Estimated); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Anxiety
Keywords: Melatonin; Lumbar medial branch block (LMBB); Anxiety; Interventional Pain; Pain Procedure
MeSH Terms: conditions — Anxiety Disorders | interventions — Melatonin; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 2 mg Melatonin (Active Comparator): To remain within the doses used for anxiolytic effects in past studies, we plan to study the effects of 2mg melatonin.
  Interventions: Drug: 2 mg Melatonin
- 10 mg Melatonin (Active Comparator): To remain within the doses used for anxiolytic effects in past studies, we plan to study the effects of 10mg melatonin.
  Interventions: Drug: 10mg Melatonin
- Sugar Pill (Placebo Comparator): To remain within the doses used for anxiolytic effects in past studies, we plan to study the effects of two different levels of melatonin versus placebo as premedication in patients undergoing a lumbar medial branch block (LMBB) procedure.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 2 mg Melatonin — 40 patients will randomly receive 2 mg melatonin
  Other Names: N-acetyl-5-methoxytripatamin
  Arms: 2 mg Melatonin
Drug: 10mg Melatonin — 40 patients will randomly receive 10 mg melatonin
  Other Names: N-acetyl-5-methoxytripatamin
  Arms: 10 mg Melatonin
Other: Placebo — 40 patients will randomly receive a placebo/sugar pill
  Other Names: Sugar Pill
  Arms: Sugar Pill

SUMMARY:
Lumbar medial branch blocks are commonly used as a diagnostic tool for facet-mediated chronic low back pain. This interventional pain procedure often occurs in the fluoroscopy suite. During this procedure, a physician inserts the needles to deliver local anesthetics such as lidocaine or bupivacaine to the nerves which innervate the lumbar facet joint. Many patients experience anxiety before and during the lumbar medial branch block procedure and require intravenous midazolam or fentanyl for sedation. Intravenous or conscious sedation requires one-to-one nursing care, monitoring, and recovery. In order to minimize the costs and time requirements of intravenous sedation, a suitable oral medication which is readily available and non-controlled would be ideal. Several randomized double-blinded, controlled trials have investigated the anxiolytic effects of melatonin before a surgery; however no studies to date have studied the anxiolytic effects of melatonin before less invasive interventional pain procedures. This study is designed to evaluate the efficacy of melatonin for reducing anxiety in patients undergoing a lumbar medial branch block procedure.

The study is a randomized, double-blinded, placebo-controlled trial with 40 patients in each group: 2 mg melatonin, 10 mg melatonin and placebo. The primary outcome is anxiety reduction in patients before undergoing the procedure. The primary outcome is measured by visual numerical rating scale for anxiety and the Amsterdam Preoperative Anxiety and Information Scale. Based on the results of previous studies, the investigators hypothesize that melatonin may reduce anxiety in patients undergoing the procedure and be a suitable alternative to intravenous sedation in the pain clinic for patients undergoing lumbar medial branch blocks.

DETAILED DESCRIPTION:
Chronic low back pain is a common disease in industrialized countries which affect patients' productivity and quality of life. Currently, the estimated yearly prevalence of chronic low back pain in United States is 5-20%. Lumbar medial branch blocks (LMBB) are commonly used as a diagnostic tool for facet mediated chronic low back pain. This interventional pain procedure often occurs in the fluoroscopy suite. During this procedure, a physician inserts the needles to deliver local anesthetics such as lidocaine or bupivacaine to the nerves which innervate the lumbar facet joint.

Many patients experience anxiety before the LMBB procedure and require intravenous midazolam or fentanyl for sedation. In fact, in a retrospective review of over 8,000 interventional fluoroscopically guided pain procedures, the highest incidence of vasovagal episodes occurred with LMBB procedures. A nurse is required to administer these medications and monitor patient's vital signs. In addition, recovery from these medications can unduly prolong the patients visit and, in the case of fentanyl, can confound the diagnostic utility of the LMBB procedure by decreasing patient's pain.

In an effort to minimize the cost of administration, monitoring, time of recovery and maximize the diagnostic utility of LMBBs, a suitable alternative is required. Several randomized, double-blinded, controlled trials investigate the anxiolytic effect of melatonin before a surgery. Several other studies and review articles describe the use of melatonin for both sedation and anxiolysis in both adults and children. However, no studies to date describe the use of melatonin for anxiolysis or sedation for interventional pain medicine procedures.

Melatonin ((N-acetyl-5-methoxytryptamine) is an over-the-counter product which patients can take to reduce anxiety before a procedure; it is a hormone produced in the pineal gland and secreted into the blood and cerebrospinal fluid. Melatonin has several functions including the regulation of circadian rhythms and regulation of the reproductive axis and antioxidant activity. Exogenous melatonin has been used to treat insomnia and jet lag.

ELIGIBILITY:
Inclusion Criteria:

* undergoing LMBB procedure
* both genders between the ages of 18-50

Exclusion Criteria:

* patients with active pregnancy (due to ionizing radiation)
* liver disease
* contraindications to LMBB procedure
* patient refusal
* localized or systemic infection
* low platelet count
* fibromyalgia
* use of sedative medications
* failure to comply with procedures
* investigator's determination that the assigned treatment is ineffective or unsafe
* appearance of unacceptable side effects in the subject

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-07; Primary Completion 2022-05 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
Change in anxiety level scores as assessed by the data collection sheet given to patients at all three time points (listed below) | Anxiety levels will be assessed at check-in time (90 minutes before procedure), immediately before procedure, and 90 minutes post-operatively.
  Comparing melatonin and placebo to see if differing levels of melatonin helps prevent or alleviate anxiety in service members undergoing an interventional pain procedure. For patients participating in the LMBB, anxiety level scores will be compared among the three time-points. Primary analysis will compare the two treatment groups versus placebo. The goal of this study is to demonstrate whether melatonin has anxiolytic effects preoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Rick Fisher, DO, Principal Investigator — United States Naval Medical Center, San Diego
Locations (2):
- United States (2):
  - Pain Medicine Center, San Diego, California
  - Naval Medical Center Portsmouth, Portsmouth, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wheeler AH. Diagnosis and management of low back pain and sciatica. Am Fam Physician. 1995 Oct;52(5):1333-41, 1347-8. PMID 7572557
- [Background] Slipman CW, Derby R, Simeone FA, et al. Slipman: Interventional Spine: An Algorithmic Approach, 1st ed. Elsevier Inc 2008.
- [Background] Wurtman R. Physiology and clinical use of melatonin. www.uptodate.com. Accessed 2/8/15.
- [Background] Cramer H, Rudolph J, Consbruch U, Kendel K. On the effects of melatonin on sleep and behavior in man. Adv Biochem Psychopharmacol. 1974;11(0):187-91. No abstract available. PMID 4367644
- [Background] Wurtman RJ, Zhdanova I. Improvement of sleep quality by melatonin. Lancet. 1995 Dec 2;346(8988):1491. doi: 10.1016/s0140-6736(95)92509-0. No abstract available. PMID 7491013
- [Background] Brzezinski A, Vangel MG, Wurtman RJ, Norrie G, Zhdanova I, Ben-Shushan A, Ford I. Effects of exogenous melatonin on sleep: a meta-analysis. Sleep Med Rev. 2005 Feb;9(1):41-50. doi: 10.1016/j.smrv.2004.06.004. PMID 15649737
- [Background] Herxheimer A, Petrie KJ. Melatonin for the prevention and treatment of jet lag. Cochrane Database Syst Rev. 2002;(2):CD001520. doi: 10.1002/14651858.CD001520. PMID 12076414
- [Background] Acil M, Basgul E, Celiker V, Karagoz AH, Demir B, Aypar U. Perioperative effects of melatonin and midazolam premedication on sedation, orientation, anxiety scores and psychomotor performance. Eur J Anaesthesiol. 2004 Jul;21(7):553-7. doi: 10.1017/s0265021504007094. PMID 15318468
- [Background] Naguib M, Samarkandi AH. The comparative dose-response effects of melatonin and midazolam for premedication of adult patients: a double-blinded, placebo-controlled study. Anesth Analg. 2000 Aug;91(2):473-9. doi: 10.1097/00000539-200008000-00046. PMID 10910871
- [Background] Caumo W, Torres F, Moreira NL Jr, Auzani JA, Monteiro CA, Londero G, Ribeiro DF, Hidalgo MP. The clinical impact of preoperative melatonin on postoperative outcomes in patients undergoing abdominal hysterectomy. Anesth Analg. 2007 Nov;105(5):1263-71, table of contents. doi: 10.1213/01.ane.0000282834.78456.90. PMID 17959953
- [Background] Ismail SA, Mowafi HA. Melatonin provides anxiolysis, enhances analgesia, decreases intraocular pressure, and promotes better operating conditions during cataract surgery under topical anesthesia. Anesth Analg. 2009 Apr;108(4):1146-51. doi: 10.1213/ane.0b013e3181907ebe. PMID 19299777
- [Background] Moerman N, van Dam FS, Muller MJ, Oosting H. The Amsterdam Preoperative Anxiety and Information Scale (APAIS). Anesth Analg. 1996 Mar;82(3):445-51. doi: 10.1097/00000539-199603000-00002. PMID 8623940
- [Background] Melatonin Monograph. http://www.naturaldatabase.com/(S(nqojvt553k2ihb45ojhbdwu1))/nd/Search.aspx?cs=CPCE&s=ND&pt=100&id=940&ds=&name=MELATONIN&searchid=17337409. Accessed 2/3/15.
- [Background] Ahmad RA, Samarkandi A, Al-Mansouri SM, Obeidan SA. Sedation characteristics of melatonin and midazolam for premedication of adult patients undergoing cataract surgery under local anesthesia. Saudi Journal of Anesthesia 2007;1(1):6.
- [Background] Bajaj P. Melatonin for anxiolysis in children. Indian J Anaesth 2009;53:504-5.
- [Background] Kucukakin, B. Modification of surgical stress response by perioperative melatonin administration. PhD Thesis for Department of Surgical Gastroenterology, University of Copenhagen,
- [Background] Kurdi MS, Patel T. The role of melatonin in anaesthesia and critical care. Indian J Anaesth. 2013 Mar;57(2):137-44. doi: 10.4103/0019-5049.111837. PMID 23825812
- [Background] Samarkandi A, Naguib M, Riad W, Thalaj A, Alotibi W, Aldammas F, Albassam A. Melatonin vs. midazolam premedication in children: a double-blind, placebo-controlled study. Eur J Anaesthesiol. 2005 Mar;22(3):189-96. doi: 10.1017/s0265021505000335. PMID 15852991
- [Background] Yousaf F, Seet E, Venkatraghavan L, Abrishami A, Chung F. Efficacy and safety of melatonin as an anxiolytic and analgesic in the perioperative period: a qualitative systematic review of randomized trials. Anesthesiology. 2010 Oct;113(4):968-76. doi: 10.1097/ALN.0b013e3181e7d626. PMID 20823763
- [Background] Andersen LP, Rosenberg J, Gogenur I. Perioperative melatonin: not ready for prime time. Br J Anaesth. 2014 Jan;112(1):7-8. doi: 10.1093/bja/aet332. No abstract available. PMID 24318695
- [Background] Capuzzo M, Zanardi B, Schiffino E, Buccoliero C, Gragnaniello D, Bianchi S, Alvisi R. Melatonin does not reduce anxiety more than placebo in the elderly undergoing surgery. Anesth Analg. 2006 Jul;103(1):121-3, table of contents. doi: 10.1213/01.ane.0000222476.62547.ed. PMID 16790638
- [Background] Pokharel K, Tripathi M, Gupta PK, Bhattarai B, Khatiwada S, Subedi A. Premedication with oral alprazolam and melatonin combination: a comparison with either alone--a randomized controlled factorial trial. Biomed Res Int. 2014;2014:356964. doi: 10.1155/2014/356964. Epub 2014 Jan 12. PMID 24527443
- [Background] Kennedy DJ, Schneider B, Casey E, Rittenberg J, Conrad B, Smuck M, Plastaras CT. Vasovagal rates in flouroscopically guided interventional procedures: a study of over 8,000 injections. Pain Med. 2013 Dec;14(12):1854-9. doi: 10.1111/pme.12241. Epub 2013 Oct 4. PMID 24118835
- [Derived] Madsen BK, Zetner D, Moller AM, Rosenberg J. Melatonin for preoperative and postoperative anxiety in adults. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD009861. doi: 10.1002/14651858.CD009861.pub3. PMID 33319916

DOCUMENTS (1):
  • Informed Consent Form (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT02415309/ICF_000.pdf